CLINICAL TRIAL: NCT05130112
Title: Impact of Airways Function After Short-term Use of High-flow Nasal Cannula Gas Therapy Evaluated by Impulse Oscillometry Systems in Stable Chronic Obstructive Pulmonary Disease Patients
Brief Title: Impact of Airways Function After HFNC Evaluated by IOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C107177
Record Dates: First submitted 2021-10-07; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: Small Airway Disorders; COPD
Keywords: high-flow nasal cannula; high nasal flow; chronic obstructive pulmonary disease (COPD); airway impedance; distal airway; peripheral airway; airway resistance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cannula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- HFNC then NC (Experimental): High flow nasal cannula for 10 min (Period 1) and nasal cannula for 10 min (Period 2) after a 4-week washout period
  Interventions: Device: high flow nasal cannula and nasal cannula
- NC then HFNC (Experimental): Nasal cannula for 10 min (Period 1) and high flow nasal cannula for 10 min (Period 2) after a 4-week washout period
  Interventions: Device: high flow nasal cannula and nasal cannula

INTERVENTIONS:
Device: high flow nasal cannula and nasal cannula — HFNC was administered using the MyAIRVO 2 device (Fisher & Paykel Healthcare, Auckland, New Zealand), which provides humidification and high-flow medical gas through an Optiflow NC interface (Fisher & Paykel Healthcare, Auckland, New Zealand) is administered for 10 min..
  NC is administered for 10 min.

SUMMARY:
In addition to pharmacological treatment, nonpharmacological treatment with high-flow nasal cannula (HFNC) may play a vital role in the treatment of patients with chronic obstructive pulmonary disease (COPD). The impulse oscillation system (IOS) is new noninvasive technique to measure the impedance of different portions of the airway with higher sensitivity than that of the conventional pulmonary function test (PFT). However, whether IOS is an appropriate technique to evaluate the efficacy of HFNC in improving the impedance of peripheral small airways in patients with COPD is unclear.

DETAILED DESCRIPTION:
Participants with stable COPD from the chest medicine outpatient department will be randomized into two groups receiving HFNC or nasal cannula (NC) for 10 min followed by a 4-week washout period and crossover alternatively. We used a novel analytical measurement technique, IOS, to detect the difference in airway impedance in the participants after the HFNC or NC interventions. All data, namely IOS parameters, transcutaneous partial pressure of carbon dioxide, peripheral oxygen saturation, body temperature, respiratory rate, pulse rate, blood pressure, and PFT results at the time of pre-HFNC, post-HFNC, pre-NC, and post-NC, were analysed using SPSS (version 25.0, IBM, Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* age of 20 to 75 years old
* diagnosis of COPD made by pulmonologist (Kuo YL) if the patient had a long-term smoking or noxious gas exposure history, typical clinical manifestations, and airflow limitation with a postbronchodilator FEV1/FVC ratio of < 0.7 in spirometry,4 and
* provision of written informed consent.

Exclusion Criteria:

* severe and unstable comorbidities or active malignancy
* history of obstructive sleep apnoea syndrome
* COPD exacerbation within the 4 weeks prior
* current use of long-term oxygen therapy or noninvasive ventilation or use within the 6 weeks prior
* cognitive impairment or a psychiatric disorder
* pregnancy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
R5 | immediately after 10 minutes of HFNC or NC
  Changes of R5
R5% | immediately after 10 minutes of HFNC or NC
  Changes of R5%
R20 | immediately after 10 minutes of HFNC or NC
  Changes of R20
R20% | immediately after 10 minutes of HFNC or NC
  Changes of R20%
Changes of R5-20 | immediately after 10 minutes of HFNC or NC
  R5-20
X5-predicted | immediately after 10 minutes of HFNC or NC
  Changes of X5-predicted
X5-predicted% | immediately after 10 minutes of HFNC or NC
  Changes of X5-predicted%
Changes of Fres | immediately after 10 minutes of HFNC or NC
  Fres
Changes of Fres% | immediately after 10 minutes of HFNC or NC
  Fres%
Changes of Ax | immediately after 10 minutes of HFNC or NC
  Ax
Ax% | immediately after 10 minutes of HFNC or NC
  Changes of Ax%

SECONDARY OUTCOMES:
TcPCO2 | immediately after 10 minutes of HFNC or NC
  Changes of TcPCO2
Body temperature | immediately after 10 minutes of HFNC or NC
  Changes of body temperature
pulse rate | immediately after 10 minutes of HFNC or NC
  Changes of pulse rate
respiratory rate | immediately after 10 minutes of HFNC or NC
  Changes of respiratory rate
both systolic and diastolic blood pressure | immediately after 10 minutes of HFNC or NC
  Changes of both systolic and diastolic blood pressure
SpO2 | immediately after 10 minutes of HFNC or NC
  Changes of SpO2
FEV1 | immediately after 10 minutes of HFNC or NC
  Changes of FEV1
FEV1% | immediately after 10 minutes of HFNC or NC
  Changes of FEV1%
FVC | immediately after 10 minutes of HFNC or NC
  Changes of FVC
FVC% | immediately after 10 minutes of HFNC or NC
  Changes of FVC%
FEV1/FVC% | immediately after 10 minutes of HFNC or NC
  Changes of FEV1/FVC%
Changes of FEV3 | immediately after 10 minutes of HFNC or NC
  FEV3
FEV3% | immediately after 10 minutes of HFNC or NC
  Changes of FEV3%
FEV3/FVC% | immediately after 10 minutes of HFNC or NC
  Changes of FEV3/FVC%
MMEF | immediately after 10 minutes of HFNC or NC
  Changes of MMEF
Changes of MMEF% | immediately after 10 minutes of HFNC or NC
  MMEF%
PEF | immediately after 10 minutes of HFNC or NC
  Changes of PEF
PEF% | immediately after 10 minutes of HFNC or NC
  Changes of PEF%

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Liang Kuo, MD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Yen-Liang Kuo, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuo YL, Chien CL, Ko HK, Lai HC, Lin TL, Lee LN, Chang CY, Shen HS, Lu CC. High-flow nasal cannula improves respiratory impedance evaluated by impulse oscillometry in chronic obstructive pulmonary disease patients: a randomised controlled trial. Sci Rep. 2022 Apr 28;12(1):6981. doi: 10.1038/s41598-022-10873-x. PMID 35484186